CLINICAL TRIAL: NCT02511379
Title: Clinical Evaluation of Systane® Balance on Corneal Staining in Indian Subjects With Dry Eye
Brief Title: Clinical Evaluation of Systane® Balance in Dry Eye Subjects
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Discontinuation of product development
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXJ821-P001 (C-13-039); CTRI/2015/10/006320 (Registry Identifier: CTRI)
Record Dates: First submitted 2015-07-28; First posted 2015-07-30 (Estimated); Results first posted 2018-09-05 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Propylene Glycol; Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Systane Balance (Experimental): Propylene Glycol 0.6% eye drops, 1 drop QID (with the last dose of each day at bedtime) in each eye for 90 days
  Interventions: Other: Propylene Glycol 0.6% eye drops

INTERVENTIONS:
Other: Propylene Glycol 0.6% eye drops
  Other Names: Systane® Balance

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Systane® Balance following 90 days of QID (4 times/day) dosing among Indian subjects with dry eye.

DETAILED DESCRIPTION:
This study was conducted in India.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent and willing and able to attend all study visits;
* Dry eye in both eyes diagnosed by an ophthalmologist;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Women of childbearing potential who are pregnant or breastfeeding;
* Any medical condition (systemic or ophthalmic) that may preclude the safe administration of test article or safe participation in the study;
* Ocular surgery or ocular trauma requiring medical or pharmacological treatment within 1 year of Screening;
* Use of topical ocular prescription or non-prescription medications, RESTASIS or topical ocular steroids within 14 days of Screening;
* Use of any artificial tears/gels/lubricants/rewetting drops within 4 hours of Screening;
* Contact lens wear within 1 week of Screening and/or unwillingness to discontinue contact lens wear for the duration of the study;
* Other protocol-specified exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-11-26 (Actual); Primary Completion 2016-06-20 (Actual); Study Completion 2016-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon Research, Ltd, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 4 study sites located in India.
Groups:
- Systane Balance: Propylene Glycol 0.6% eye drops, 1 drop QID (4 times/day) (with the last dose of each day at bedtime) in each eye for 90 days
Period: Overall Study
Arm/Group | Systane Balance
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Systane Balance
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Corneal Staining Total Score
Description: The type (severity) of staining was assessed for each of the 5 regions of the cornea (central, inferior, temporal, superior, and nasal) and graded on a 4-point scale, where 0 = Normal (No staining) and 3 = Severe (Numerous coalescent macropunctate areas and/or patches). The scores of the 5 regions were summed to obtain a corneal staining total score for each eye (minimum 0, maximum 15).
Time Frame: Baseline (Day 0), Day 45, Day 90
Population: Analysis includes all participants with data present. Analysis was based on the eye with the higher corneal staining total score at screening or the right eye when both eyes have same corneal staining total score at screening, as observed.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Systane Balance
Number analyzed (Participants) | 14
units on a scale
  Change from baseline at Day 45 | -3.1 [-8 to 1]
  Change from baseline at Day 90: number analyzed (Participants) | 13
  Change from baseline at Day 90 | -4.8 [-11 to -1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of participation, an average of 90 days.
Arm/Group | Systane Balance
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes